CLINICAL TRIAL: NCT02665481
Title: Remediating Age Related Cognitive Decline: Mindfulness-Based Stress Reduction and Exercise
Brief Title: Mindfulness-Based Stress Reduction, Health Education and Exercise
Acronym: MEDEX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: University of California, San Diego (Other); National Institutes of Health (NIH) (NIH); National Institute on Aging (NIA) (NIH); National Center for Complementary and Integrative Health (NCCIH) (NIH); The Brain Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 201410093; 1R01AG049369-01 (NIH)
Record Dates: First submitted 2016-01-12; First posted 2016-01-27 (Estimated); Results first posted 2022-09-28 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Age-related Cognitive Decline
Keywords: Exercise; Mindfulness; Education; Elderly
MeSH Terms: conditions — Motor Activity | interventions — Mindfulness-Based Stress Reduction; Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- MBSR (Experimental): Mindfulness-Based Stress Reduction consists of a brief introductory meeting, eight weekly 2.5-hour classes, and a retreat, followed by monthly booster sessions for approximately 15 months. Content includes instruction in mindfulness meditation practices, gentle mindful movement, and exercises to enhance mindfulness in everyday life.
  Interventions: Behavioral: MBSR
- Exercise (Experimental): The exercise protocol is optimal for improving aerobic fitness and insulin sensitivity in older adults, as well as improving strength and balance and reducing indices of frailty.It consists of classes twice weekly for 6 months, building up to 1.5 hr, under the direct supervision of trained exercise instructors, followed by once weekly classes for 12 months.
  Interventions: Behavioral: Exercise
- MBSR + Exercise (Experimental): This condition will receive both MBSR and exercise as described above. Participants in this condition will come in once weekly to receive MBSR and twice weekly to receive exercise classes, with at-home exercise the other two days as well as daily, at-home mindfulness practice. After the initial classes participants will also attend additional weekly or monthly sessions until completion of the study.
  Note that at each site a pilot group is undergoing MBSR + Exercise (not randomized, separate from the RCT).
  Interventions: Behavioral: MBSR; Behavioral: Exercise
- Health Education (Active Comparator): Health Education is a group-based intervention that increases health-related knowledge and action. Health Education improves chronic disease management.Health Education consists of ten weekly 2.5-hour classes, followed by monthly classes for approximately 15 months.
  Interventions: Behavioral: Health Education

INTERVENTIONS:
Behavioral: MBSR
  Other Names: Mindfulness-Based Stress Reduction
  Arms: MBSR; MBSR + Exercise
Behavioral: Exercise
  Other Names: Multi-component intensity-based exercise
  Arms: Exercise; MBSR + Exercise
Behavioral: Health Education
  Arms: Health Education

SUMMARY:
The purpose of this research is to examine the effects of four interventions on age-related cognitive decline in healthy older adults. The investigators will examine the effects of Mindfulness Based Stress Reduction (MBSR) psychotherapy, multi-component intensity-based aerobic exercise, and their combination, compared to a discussion group.

DETAILED DESCRIPTION:
MBSR teaches mindfulness, or the focusing of attention and awareness, through various meditation techniques. Mindfulness meditation practices appear to produce neurocircuitry changes that are the reverse of those seen in age-related cognitive decline. It is widely available, acceptable to older people, and carries minimal risk of side effects or adverse events. Exercise - specifically, intense, multi-component exercise - also appears to affect brain structure and function and improve cognitive performance.

The investigators will randomize 580 non-demented healthy adults aged 65 to 84 to one of four conditions: MBSR alone, exercise alone, MBSR + exercise, or a health education discussion group control condition.

The study will consist of a 6-month acute intervention phase with weekly visits followed by a 12-month maintenance phase with weekly or monthly visits and other prompts to maintain intervention behaviors.

Assessments include cognitive tests, biomarkers, neuroimaging assessments, functional assessments to examine real-world benefits of the interventions, and other behavioral assessments to characterize participants and pave the way for further exploratory analyses.

ELIGIBILITY:
Inclusion Criteria:

* Community-living men and women age 65 to 84.
* Self-reported cognitive complaints that are a normal part of aging.
* No current meditation practice nor prior training in it.
* Sedentary.

Exclusion Criteria:

* Known diagnosis of dementia, mild cognitive impairment, other clinical neurodegenerative illness (e.g., Parkinson's disease, cerebrovascular disease), psychotic disorder, or any unstable psychiatric condition.
* Medical conditions that suggest shortened lifespan, such as metastatic cancer; or would prohibit safe participation in the interventions, including cardiovascular disease or musculoskeletal conditions; or would interfere with the assessments, such as taking medications for diabetes or ferromagnetic metal/bridgework that would interfere with MRI signal.
* IQ <70 as estimated by the Wechsler Test of Adult Reading
* Sensory impairment (language, hearing, or visual) that would prevent participation.
* Alcohol abuse within 6 months.
* Current illicit drug use.
* Concurrent cognitive training, such as brain-training software, or other interventions expected to affect neuroplasticity.
* Medications that interfere with measurements, including cancer chemotherapy, glucocorticoids, and interferon.
* Inability to cooperate with protocol.

Ages: 65 Years to 84 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 585 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2020-06 (Actual); Study Completion 2021-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric J Lenze, MD, Principal Investigator — Washington University School of Medicine
Locations (2):
- United States (2):
  - University of California San Diego, San Diego, California
  - Washington University School of Medicine, St Louis, Missouri

IPD SHARING:
Plan to Share IPD: Yes
A cleaned, complete, and de-identified copy of the final data set including administrative and technical metadata records will be made available for release upon request to qualified investigators.

REFERENCES:
- [Derived] Lenze EJ, Voegtle M, Miller JP, Ances BM, Balota DA, Barch D, Depp CA, Diniz BS, Eyler LT, Foster ER, Gettinger TR, Head D, Hershey T, Klein S, Nichols JF, Nicol GE, Nishino T, Patterson BW, Rodebaugh TL, Schweiger J, Shimony JS, Sinacore DR, Snyder AZ, Tate S, Twamley EW, Wing D, Wu GF, Yang L, Yingling MD, Wetherell JL. Effects of Mindfulness Training and Exercise on Cognitive Function in Older Adults: A Randomized Clinical Trial. JAMA. 2022 Dec 13;328(22):2218-2229. doi: 10.1001/jama.2022.21680. PMID 36511926
- See also: Visit the Healthy Mind Lab for more information about the MEDEX study and our other areas of research. STL: http://healthymind.wustl.edu/medex UCSD: http://www.medexstudy.com/ — http://healthymind.wustl.edu/medex

RESULTS

PARTICIPANT FLOW:
Groups:
- MBSR: Mindfulness-Based Stress Reduction consists of a brief introductory meeting, eight weekly 2.5-hour classes, and a retreat, followed by monthly booster sessions for approximately 15 months. Content includes instruction in mindfulness meditation practices, gentle mindful movement, and exercises to enhance mindfulness in everyday life.
  MBSR
- Exercise: The exercise protocol is optimal for improving aerobic fitness and insulin sensitivity in older adults, as well as improving strength and balance and reducing indices of frailty.It consists of classes twice weekly for 6 months, building up to 1.5 hr, under the direct supervision of trained exercise instructors, followed by once weekly classes for 12 months.
  Exercise
- MBSR + Exercise: This condition will receive both MBSR and exercise as described above. Participants in this condition will come in once weekly to receive MBSR and twice weekly to receive exercise classes, with at-home exercise the other two days as well as daily, at-home mindfulness practice. After the initial classes participants will also attend additional weekly or monthly sessions until completion of the study.
  Note that at each site a pilot group is undergoing MBSR + Exercise (not randomized, separate from the RCT).
  MBSR
  Exercise
- Health Education: Health Education is a group-based intervention that increases health-related knowledge and action. Health Education improves chronic disease management.Health Education consists of ten weekly 2.5-hour classes, followed by monthly classes for approximately 15 months.
  Health Education
Period: Overall Study
Arm/Group | MBSR | Exercise | MBSR + Exercise | Health Education
Started | 150 | 138 | 144 | 153
Completed | 139 | 119 | 106 | 111
Not Completed | 11 | 19 | 38 | 42

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MBSR | Exercise | MBSR + Exercise | Health Education | Total
Number analyzed (Participants) | 150 | 138 | 144 | 153 | 585
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.2 (4.2) | 71.1 (4.9) | 72.4 (5.3) | 71.1 (4.6) | 71.5 (4.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 108 | 108 | 102 | 106 | 424
  Male | 42 | 30 | 42 | 47 | 161
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian/Alaska Native | 0 | 1 | 1 | 0 | 2
  Asian | 3 | 9 | 10 | 5 | 27
  Black or African American | 18 | 14 | 18 | 19 | 69
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  White | 127 | 109 | 112 | 129 | 477
  More than one race | 1 | 0 | 3 | 0 | 4
  Unknown/not reported | 1 | 5 | 0 | 0 | 6
  Hispanic | 7 | 9 | 14 | 9 | 39
Current smoker [Count of Participants; unit: Participants] | 4 | 1 | 0 | 5 | 10
Years of education [Mean (Standard Deviation); unit: years] | 16.0 (2.2) | 16.6 (2.2) | 16.0 (2.3) | 16.1 (2.1) | 16.2 (2.2)
APOE 4 positive [Count of Participants; unit: Participants] — ApoE is a gene which can dramatically increase your risk for Alzheimer's. Patients who test positive for the apolipoprotein E4 (ApoE4) gene demonstrate an increased chance of Alzheimer's disease.
  Participants | 49 | 44 | 37 | 44 | 174
CIRS-G [Mean (Standard Deviation); unit: units on a scale] — The Cumulative Illness Rating Scale for Geriatrics (CIRS-G) is a 14-item scale that assesses overall health. A total score is reported with a range of 0 to 56, where a higher score represents worse overall health.
  units on a scale | 6.7 (2.9) | 6.7 (2.8) | 6.9 (2.8) | 6.7 (3.0) | 6.8 (2.9)
CEI [Mean (Standard Deviation); unit: units on a scale] — The Credibility and Expectations Questionnaire (CEI) assessed subjective beliefs that the intervention is credible (will work). Participants also indicated their expectations that the assigned intervention would improve their condition (i.e. cognition). This questionnaire was given only after the first class. The credibility portion of the questionnaire consisted of four items (total score from 0 to 40), with a higher score representing more credibility. The expectation portion of the questionnaire consisted of one item, a percentage from 0% to 100% (higher: expect greater improvement).
  units on a scale
    Credibility | 30.1 (6.8) | 33.5 (5.8) | 32.9 (6.4) | 26.6 (7.4) | 30.6 (7.2)
    Improvement | 59.4 (24.2) | 61.9 (23.5) | 68.4 (23.0) | 56.1 (22.5) | 61.3 (23.7)
Body Mass Index (BMI) Class [Count of Participants; unit: Participants] — Body mass index or BMI is a statistical index using a person's weight and height to get an estimate of body fat in persons of any age.
  Participants
    Normal (16-24.9 kg/m^2) | 57 | 34 | 35 | 47 | 173
    Overweight (25-29.9 kg/m^2) | 51 | 51 | 63 | 54 | 219
    Obese (30.0+ kg/m^2) | 42 | 53 | 46 | 52 | 193
WTAR [Mean (Standard Deviation); unit: units on a scale] — The Wechsler Test of Adult Reading (WTAR) instrument is used to gain an estimate of IQ. Participants read 50 words from a page and were scored on correct pronunciation. Those with a standard score less than 70 were not eligible to participate in the study. The minimum raw score is 0 and the maximum raw score is 50. The standard score ranges from 52 to 128. The higher the score, the higher the estimated IQ.
  units on a scale
    Raw score | 41.5 (7.1) | 41.9 (6.7) | 41.4 (7.0) | 40.6 (6.9) | 41.3 (6.9)
    Standard score | 113.6 (10.6) | 114.1 (10.2) | 113.4 (10.4) | 112.2 (10.3) | 113.3 (10.4)
SPPB modified score [Mean (Standard Deviation); unit: units on a scale] — The Short Physical Performance Battery (SPPB) measures gait speed, chair stand and balance. It is used as a tool for detecting disability and can help monitor the function in older adults. A total score was computed by summing the scores of gait speed, chair stand, and balance. The total score has a range from 1 to 12 where a higher score indicates higher functioning. All balance testing was measured using BtrackS balance tracking system, a computerized force platform provided a more objective and detailed assessment of balance than observation alone.
  units on a scale | 8.8 (1.8) | 8.7 (1.9) | 9.0 (2.0) | 8.8 (2.0) | 8.8 (1.9)
Paragraph recall [Mean (Standard Deviation); unit: units on a scale] — The Paragraph Recall task involves having the participant listen to two stories and then asking the participant to remember as many of the paragraph elements as possible. Each story has 44 elements. Therefore, the range is 0 to 88 for both the immediate recall task and the delayed recall task. The task is used to quantify memory performance. The greater the score, the higher the memory performance.
  units on a scale
    Immediate positive total | 43.0 (10.7) | 43.4 (10.2) | 41.9 (10.8) | 42.6 (9.8) | 42.7 (10.4)
    Delayed positive total | 36.4 (12.0) | 37.5 (10.8) | 35.8 (11.3) | 36.7 (10.1) | 36.6 (11.1)
Word list [Mean (Standard Deviation); unit: units on a scale] — The Word List Learning and Recall tasks involve the participant recalling as many words as possible from a list containing 16 words. For the Learning task, the participant will try to recall as many words as possible for 4 trials. Therefore, the total score ranges from 0 to 64. The Recall task occurs 20 minutes following the Learning task, and again has the participant recall as many words as possible from the list. It has a range of 0 to 16. In both the Learning and Recall tasks, the higher the score, the better the outcome.
  units on a scale
    Learning | 32.4 (7.4) | 31.3 (7.3) | 31.2 (7.6) | 31.1 (7.4) | 31.5 (7.4)
    Recall | 6.9 (3.1) | 7.1 (3.2) | 6.6 (3.0) | 6.5 (3.2) | 6.8 (3.1)
Neuro-QoL cognitive function score [Mean (Standard Deviation); unit: units on a scale] — The Quality of Life in Neurological Disorders (NQoL) Cognitive Function Scale is an 18-item self-report measure that assesses the health-related quality of life of adults. The total score ranges from 18 to 90 where a higher score represents a better outcome.
  units on a scale | 62.4 (12.6) | 63.2 (12.1) | 65.5 (11.4) | 63.3 (11.4) | 63.6 (11.9)
OTDL-R [Mean (Standard Deviation); unit: units on a scale] — The Revised Observed Tasks of Daily Living (OTDL-R) is a performance-based test of everyday problem-solving. Subjects completed tasks testing medication use (following medicine label directions, and completing a patient record form); telephone use (finding and dialing a number from the yellow pages); and financial management (making change with coins and bills, and balancing a checkbook). The scores were summed with the total score having a range from 0 to 28. The higher the score, the more likely the participant is able to complete everyday activities.
  units on a scale | 20.7 (3.2) | 20.4 (3.5) | 20.3 (3.5) | 20.2 (3.7) | 20.4 (3.5)
CAMS-R [Mean (Standard Deviation); unit: units on a scale] — The Cognitive and Affective Mindfulness Scale-Revised (CAMS-R) is a brief 12-item self-report measure of mindfulness with items written in everyday language. Scores on the scale are summed with a range of 0 to 48. Higher values reflect greater mindful qualities.
  units on a scale | 38.1 (6.2) | 37.0 (5.6) | 37.8 (5.9) | 36.7 (5.6) | 37.4 (5.9)
NIH Toolbox Fluid Cognition Composite Score [Mean (Standard Deviation); unit: units on a scale] — This score was derived from averaging the standard scores of the Flanker, Dimensional Change Card Sort, Picture Sequence Memory, List Sorting and Pattern Comparison tasks, and then deriving standard scores based on this new distribution. An uncorrected standard score at or near 100 indicates ability that is average compared with others nationally. A standard score of around 85 suggests significantly below-average fluid cognitive ability. The population mean is 100 with a standard deviation of 15. This scale does not have a full scale range.
  units on a scale | 92.0 (8.7) | 92.0 (10.0) | 91.4 (8.4) | 91.5 (9.1) | 91.7 (9.0)
Cortisol AUC [Mean (Standard Deviation); unit: mcg*min/mL] | 5580 (2471) | 5703 (2606) | 6565 (2950) | 5749 (2500) | 5892 (2653)
Insulin sensitivity [Mean (Standard Deviation); unit: units on a scale] — Homeostasis Model Assessment of Insulin Resistance (HOMA-IR) measures how insulin resistant (IR) an individual is with a higher HOMA-IR indicating greater IR. HOMA-IR is computed using the fasting glucose and insulin values of an OGTT. The Oral Glucose Insulin Sensitivity (OGIS) index assesses insulin sensitivity using the insulin and glucose values obtained at the 0, 90, and 120-time points from a 2-hr OGTT. The higher the OGIS index, the more insulin sensitive an individual is. An OGIS of 302 (+/- 17) suggests impaired glucose tolerance. A HOMA-IR less than 1.0 indicates insulin sensitivity.
  units on a scale
    HOMA-IR | 2.5 (1.7) | 3.0 (2.2) | 3.0 (2.1) | 3.1 (2.3) | 2.9 (2.1)
    OGIS (ml*min-1*m-2) | 352 (61) | 344 (63) | 348 (67) | 346 (67) | 348 (64)

OUTCOME MEASURES:

1. Primary Outcome: Memory Composite Score
Description: The memory composite variable consists of the list recall, paragraph recall, and picture sequence memory tasks. For each memory variable, a z score is computed for each participant [(participant score - mean)/standard deviation]. Then the composite memory variable is created by averaging the z scores. The higher the z-score, the better the outcome. A Z-score of 0 represents the population mean.
Time Frame: Month 0, Month 3, Month 6, and Month 18
Population: modified Intent-to-Treat, which includes all participants that received at least one dose of the intervention.
Measure: Least Squares Mean (Standard Error); unit: Z-score
Groups:
- MBSR Positive: This group consists of participants that received the MBSR intervention.
- MBSR Negative: This group consists of participants that did not receive the MBSR intervention.
- Exercise Positive: This group consists of participants that received the Exercise intervention.
- Exercise Negative: This group consists of participants that did not receive the Exercise intervention.
Arm/Group | MBSR Positive | MBSR Negative | Exercise Positive | Exercise Negative
Number analyzed (Participants) | 294 | 291 | 282 | 303
Z-score
  Month 0 | -0.11 (0.06) | -0.14 (0.06) | -0.13 (0.06) | -0.12 (0.06)
  Month 3 | 0.07 (0.06) | 0.04 (0.06) | 0.04 (0.06) | 0.06 (0.06)
  Month 6 | 0.33 (0.06) | 0.34 (0.06) | 0.36 (0.07) | 0.30 (0.06)
  Month 18 | 0.50 (0.06) | 0.39 (0.06) | 0.42 (0.07) | 0.47 (0.06)
Statistical Analysis 1: Comparison: MBSR Positive vs MBSR Negative; Time x MBSR (Month 0 and Month 6); Test type: Superiority; p = 0.50, Marginal Model; Mean Difference (Final Values) = -0.04, 95% CI 2-sided [-0.15 to 0.07]
Statistical Analysis 2: Comparison: MBSR Positive vs MBSR Negative; Time x MBSR (Month 0 and Month 18); Test type: Superiority; p = 0.18, Marginal Model; Mean Difference (Final Values) = 0.08, 95% CI 2-sided [-0.04 to 0.19]
Statistical Analysis 3: Comparison: Exercise Positive vs Exercise Negative; Time x Exercise (Month 0 and Month 6); Test type: Superiority; p = 0.23, Marginal Model; Mean Difference (Final Values) = 0.07, 95% CI 2-sided [-0.04 to 0.17]
Statistical Analysis 4: Comparison: Exercise Positive vs Exercise Negative; Time x Exercise (Month 0 and Month 18); Test type: Superiority; p = 0.47, Marginal Model; Mean Difference (Final Values) = -0.04, 95% CI 2-sided [-0.15 to 0.07]

2. Primary Outcome: Cognitive Control Composite Score
Description: The cognitive control composite variable uses the CVOE, SART, Color Word Interference, flanker, dimensional change card sort, and list-sorting tasks. For each cognitive variable, a z score is computed for each participant [(participant score - mean)/standard deviation]. Then the composite cognitive control variable is created by averaging the z scores. The higher the z-score, the better the outcome. A Z-score of 0 represents the population mean.
Time Frame: Month 0, Month 3, Month 6, Month 18
Population: modified Intent-to-Treat, which includes all participants that received at least one dose of the intervention.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | MBSR Positive | MBSR Negative | Exercise Positive | Exercise Negative
Number analyzed (Participants) | 294 | 291 | 282 | 303
score on a scale
  Month 0 | 0.09 (0.06) | -0.01 (0.06) | 0.05 (0.06) | 0.03 (0.06)
  Month 3 | 0.26 (0.06) | 0.21 (0.06) | 0.26 (0.06) | 0.21 (0.06)
  Month 6 | 0.48 (0.06) | 0.30 (0.06) | 0.44 (0.06) | 0.35 (0.06)
  Month 18 | 0.36 (0.06) | 0.30 (0.06) | 0.33 (0.06) | 0.32 (0.06)
Statistical Analysis 1: Comparison: MBSR Positive vs MBSR Negative; Time x MBSR (Month 0 and Month 6); Test type: Superiority; p = 0.12, Marginal Model; Mean Difference (Final Values) = 0.08, 95% CI 2-sided [-0.02 to 0.19]
Statistical Analysis 2: Comparison: MBSR Positive vs MBSR Negative; Time x MBSR (Month 0 and Month 18); Test type: Superiority; p = 0.44, Marginal Model; Mean Difference (Final Values) = -0.04, 95% CI 2-sided [-0.15 to 0.07]
Statistical Analysis 3: Comparison: Exercise Positive vs Exercise Negative; Time x Exercise (Month 0 and Month 6); Test type: Superiority; p = 0.17, Marginal Model; Mean Difference (Final Values) = 0.07, 95% CI 2-sided [-0.03 to 0.18]
Statistical Analysis 4: Comparison: Exercise Positive vs Exercise Negative; Time x Exercise (Month 0 and Month 18); Test type: Superiority; p = 0.93, Marginal Model; Mean Difference (Final Values) = -0.01, 95% CI 2-sided [-0.12 to 0.11]

3. Secondary Outcome: Hippocampal Volume
Description: The hippocampal volume is derived from structural MRI high-resolution T1-weighted images.
Time Frame: Month 0, Month 6, Month 18
Population: modified Intent-to-Treat, which includes all participants that received at least one dose of the intervention.
Measure: Least Squares Mean (Standard Error); unit: millimeters^3
Arm/Group | MBSR Positive | MBSR Negative | Exercise Positive | Exercise Negative
Number analyzed (Participants) | 274 | 268 | 253 | 289
millimeters^3
  Month 0 | 3680 (21) | 3618 (22) | 3641 (22) | 3656 (21)
  Month 6 | 3659 (21) | 3600 (22) | 3624 (22) | 3636 (21)
  Month 18 | 3613 (21) | 3571 (22) | 3581 (22) | 3602 (21)
Statistical Analysis 1: Comparison: MBSR Positive vs MBSR Negative; Time x MBSR (Month 0 and Month 6); Test type: Superiority; p = 0.53, Marginal Model; Mean Difference (Final Values) = -3.46, 95% CI 2-sided [-14.27 to 7.34]
Statistical Analysis 2: Comparison: MBSR Positive vs MBSR Negative; Time x MBSR (Month 0 and Month 18); Test type: Superiority; p = 0.004, Marginal Model; Mean Difference (Final Values) = -20.16, 95% CI 2-sided [-33.88 to -6.44]
Statistical Analysis 3: Comparison: Exercise Positive vs Exercise Negative; Time x Exercise (Month 0 and Month 6); Test type: Superiority; p = 0.58, Marginal Model; Mean Difference (Final Values) = 3.04, 95% CI 2-sided [-7.76 to 13.85]
Statistical Analysis 4: Comparison: Exercise Positive vs Exercise Negative; Time x Exercise (Month 0 and Month 18); Test type: Superiority; p = 0.37, Marginal Model; Mean Difference (Final Values) = -6.26, 95% CI 2-sided [-19.98 to 7.46]

4. Secondary Outcome: DLPFC Surface Area
Description: The Dorsal Lateral Pre-Frontal Cortex (DLPFC) surface area is derived from structural MRI high-resolution T1-weighted images.
Time Frame: Month 0, Month 6, Month 18
Population: modified Intent-to-Treat, which includes all participants that received at least one dose of the intervention.
Measure: Least Squares Mean (Standard Error); unit: millimeters^2
Arm/Group | MBSR Positive | MBSR Negative | Exercise Positive | Exercise Negative
Number analyzed (Participants) | 274 | 268 | 253 | 289
millimeters^2
  Month 0 | 12295 (80) | 12228 (82) | 12238 (84) | 12285 (78)
  Month 6 | 12296 (80) | 12207 (82) | 12220 (84) | 12284 (78)
  Month 18 | 12299 (80) | 12208 (83) | 12240 (84) | 12266 (78)
Statistical Analysis 1: Comparison: MBSR Positive vs MBSR Negative; Time x MBSR (Month 0 and Month 6); Test type: Superiority; p = 0.33, Marginal Model; Mean Difference (Final Values) = 22.71, 95% CI 2-sided [-22.95 to 68.36]
Statistical Analysis 2: Comparison: MBSR Positive vs MBSR Negative; Time x MBSR (Month 0 and Month 18); Test type: Superiority; p = 0.31, Marginal Model; Mean Difference (Final Values) = 25.35, 95% CI 2-sided [-23.18 to 73.88]
Statistical Analysis 3: Comparison: Exercise Positive vs Exercise Negative; Time x Exercise (Month 0 and Month 6); Test type: Superiority; p = 0.46, Marginal Model; Mean Difference (Final Values) = -17.18, 95% CI 2-sided [-62.83 to 28.48]
Statistical Analysis 4: Comparison: Exercise Positive vs Exercise Negative; Time x Exercise (Month 0 and Month 18); Test type: Superiority; p = 0.39, Marginal Model; Mean Difference (Final Values) = 21.11, 95% CI 2-sided [-27.41 to 69.64]

5. Secondary Outcome: DLPFC Cortical Thickness
Description: The Dorsal Lateral Pre-Frontal Cortex Cortical Thickness is derived from structural MRI high-resolution T1-weighted images.
Time Frame: Month 0, Month 6, and Month 18
Population: modified Intent-to-Treat, which includes all participants that received at least one dose of the intervention.
Measure: Least Squares Mean (Standard Error); unit: millimeters
Arm/Group | MBSR Positive | MBSR Negative | Exercise Positive | Exercise Negative
Number analyzed (Participants) | 274 | 268 | 253 | 289
millimeters
  Month 0 | 2.77 (0.01) | 2.77 (0.01) | 2.77 (0.01) | 2.77 (0.01)
  Month 6 | 2.76 (0.01) | 2.76 (0.01) | 2.76 (0.01) | 2.75 (0.01)
  Month 18 | 2.74 (0.01) | 2.75 (0.01) | 2.74 (0.01) | 2.75 (0.01)
Statistical Analysis 1: Comparison: MBSR Positive vs MBSR Negative; Time x MBSR (Month 0 and Month 6); Test type: Superiority; p = 0.37, Marginal Model; Mean Difference (Final Values) = -0.01, 95% CI 2-sided [-0.02 to 0.01]
Statistical Analysis 2: Comparison: MBSR Positive vs MBSR Negative; Time x MBSR (Month 0 and Month 18); Test type: Superiority; p = 0.10, Marginal Model; Mean Difference (Final Values) = -0.01, 95% CI 2-sided [-0.02 to 0.00]
Statistical Analysis 3: Comparison: Exercise Positive vs Exercise Negative; Time x Exercise (Month 0 and Month 6); Test type: Superiority; p = 0.21, Marginal Model; Mean Difference (Final Values) = 0.01, 95% CI 2-sided [-0.004 to 0.02]
Statistical Analysis 4: Comparison: Exercise Positive vs Exercise Negative; Time x Exercise (Month 0 and Month 18); Test type: Superiority; p = 0.09, Marginal Model; Mean Difference (Final Values) = -0.01, 95% CI 2-sided [-0.02 to 0.00]

6. Secondary Outcome: OTDL (Observed Tasks of Daily Living).
Description: The Revised Observed Tasks of Daily Living (OTDL-R) is a performance-based test of everyday problem-solving. Subjects completed tasks testing medication use (following medicine label directions, and completing a patient record form); telephone use (finding and dialing a number from the yellow pages); and financial management (making change with coins and bills, and balancing a checkbook). The scores were summed with the total score having a range from 0 to 28. The higher the score, the more likely the participant is able to complete everyday activities.
Time Frame: Month 0, Month 6, Month 18
Population: modified Intent-to-Treat, which includes all participants that received at least one dose of the intervention.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | MBSR Positive | MBSR Negative | Exercise Positive | Exercise Negative
Number analyzed (Participants) | 294 | 291 | 282 | 303
score on a scale
  Month 0 | 20.5 (0.2) | 20.2 (0.2) | 20.3 (0.2) | 20.3 (0.2)
  Month 6 | 21.7 (0.2) | 21.2 (0.2) | 21.3 (0.2) | 21.6 (0.2)
  Month 18 | 22.5 (0.2) | 22.2 (0.2) | 22.3 (0.2) | 22.3 (0.2)
Statistical Analysis 1: Comparison: MBSR Positive vs MBSR Negative; Time x MBSR (Month 0 and Month 6); Test type: Superiority; p = 0.57, Marginal Model; Mean Difference (Final Values) = 0.16, 95% CI 2-sided [-0.38 to 0.69]
Statistical Analysis 2: Comparison: MBSR Positive vs MBSR Negative; Time x MBSR (Month 0 and Month 18); Test type: Superiority; p = 0.96, Marginal Model; Mean Difference (Final Values) = -0.01, 95% CI 2-sided [-0.58 to 0.55]
Statistical Analysis 3: Comparison: Exercise Positive vs Exercise Negative; Time x Exercise (Month 0 and Month 6); Test type: Superiority; p = 0.37, Marginal Model; Mean Difference (Final Values) = -0.24, 95% CI 2-sided [-0.78 to 0.29]
Statistical Analysis 4: Comparison: Exercise Positive vs Exercise Negative; Time x Exercise (Month 0 and Month 18); Test type: Superiority; p = 0.99, Marginal Model; Mean Difference (Final Values) = -0.003, 95% CI 2-sided [-0.57 to 0.57]

7. Secondary Outcome: Quality of Life in Neurological Disorders Cognitive Function Scale (NQoL).
Description: The Quality of Life in Neurological Disorders (NQoL) Cognitive Function Scale is an 18-item self-report measure that assesses the health-related quality of life of adults. The total score ranges from 18 to 90 where a higher score represents a better outcome.
Time Frame: Month 0, Month 3, Month 6, Month 18
Population: modified Intent-to-Treat, which includes all participants that received at least one dose of the intervention.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | MBSR Positive | MBSR Negative | Exercise Positive | Exercise Negative
Number analyzed (Participants) | 294 | 291 | 282 | 303
score on a scale
  Month 0 | 64.1 (0.7) | 63.0 (0.7) | 64.4 (0.7) | 62.8 (0.7)
  Month 3 | 66.8 (0.7) | 66.0 (0.7) | 67.0 (0.7) | 65.8 (0.7)
  Month 6 | 68.3 (0.7) | 66.3 (0.7) | 67.8 (0.7) | 66.8 (0.7)
  Month 18 | 70.0 (0.7) | 67.7 (0.7) | 69.9 (0.8) | 67.8 (0.7)
Statistical Analysis 1: Comparison: MBSR Positive vs MBSR Negative; Time x MBSR (Month 0 and Month 6); Test type: Superiority; p = 0.19, Marginal Model; Mean Difference (Final Values) = 0.93, 95% CI 2-sided [-0.47 to 2.33]
Statistical Analysis 2: Comparison: MBSR Positive vs MBSR Negative; Time x MBSR (Month 0 and Month 18); Test type: Superiority; p = 0.09, Marginal Model; Mean Difference (Final Values) = 1.29, 95% CI 2-sided [-0.19 to 2.77]
Statistical Analysis 3: Comparison: Exercise Positive vs Exercise Negative; Time x Exercise (Month 0 and Month 6); Test type: Superiority; p = 0.42, Marginal Model; Mean Difference (Final Values) = -0.57, 95% CI 2-sided [-1.97 to 0.83]
Statistical Analysis 4: Comparison: Exercise Positive vs Exercise Negative; Time x Exercise (Month 0 and Month 18); Test type: Superiority; p = 0.54, Marginal Model; Mean Difference (Final Values) = 0.47, 95% CI 2-sided [-1.01 to 1.94]

ADVERSE EVENTS:
Time Frame: The adverse events and serious adverse events were collected over a period of 18 months.
Arm/Group | MBSR | Exercise | MBSR + Exercise | Health Education
All-Cause Mortality (participants affected / at risk) | 1/150 | 0/138 | 0/144 | 0/153
Serious Adverse Events (participants affected / at risk) | 18/150 | 16/138 | 14/144 | 5/153
Other Adverse Events (participants affected / at risk) | 0/150 | 0/138 | 0/144 | 0/153
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MBSR (N=150) | Exercise (N=138) | MBSR + Exercise (N=144) | Health Education (N=153)
Injury (General disorders) | 0 (0) | 3 (3) | 3 (3) | 0 (0)
Cardiovascular Event (General disorders) | 2 (2) | 4 (4) | 2 (2) | 1 (1)
Tumor/Cancer (General disorders) | 4 (4) | 0 (0) | 2 (2) | 0 (0)
Bowel Obstruction (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Asthma (Syncope) (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Blood Infection (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Ocular Migraine with Aphasia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Viral Infection (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Shingles/Urinary Tract Infection (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Leg Infection (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary Embolism (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Kidney Stone (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Inflammatory Myopathy (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neck Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Transient Ischemic Attack (TIA) (General disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Laminectomy (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Bronchitis (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Knee Replacement Surgery (General disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hip Replacement Surgery (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Enlarged Prostate (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Kidney Failure (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
High Blood Pressure (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Death (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-04-10): https://cdn.clinicaltrials.gov/large-docs/81/NCT02665481/Prot_000.pdf
  • Statistical Analysis Plan (2022-05-01): https://cdn.clinicaltrials.gov/large-docs/81/NCT02665481/SAP_001.pdf